CLINICAL TRIAL: NCT00439751
Title: A Randomized Comparison of Immediate Versus Deferred Androgen Deprivation Therapy Using Goserelin for Recurrent Prostate Cancer After Radical Radiotherapy.
Brief Title: Immediate Versus Deferred Androgen Deprivation Therapy,Goserelin for Recurrent Prostate Cancer After Radical Radiotherapy
Acronym: ELAAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-P1
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2015-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen Deprivation Therapy; Recurrence; Biochemical Failure; Goserelin
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate ADT (Other)
  Interventions: Drug: Goserelin Acetate
- Deferred ADT (Other)
  Interventions: Drug: Goserelin Acetate

INTERVENTIONS:
Drug: Goserelin Acetate — Continuous goserelin, 12 week (10.8 mg) depot, will be used as ADT for both study arms. It is supplied as a sterile syringe for subcutaneous use.
  Other Names: Zoladex®; Zoladex® LA

SUMMARY:
This is a prospective, multicentre, open-labelled, randomized controlled trial comparing the efficacy of immediate versus deferred androgen deprivation therapy (ADT) using goserelin (Zoladex®) in men with recurrent prostate cancer after radical radiotherapy.

1100 patients will be accrued from participating Canadian Urological Oncology Group sites in an estimated time of 3 years. First analysis is planned for 7 years after study recruitment is completed.

DETAILED DESCRIPTION:
Recurrent prostate cancer after radical radiation therapy is a common problem with often a long interval from biochemical failure to the time of symptomatic relapse. Androgen deprivation therapy (ADT) is the most commonly used intervention following radiation failure and currently is often started immediately after the recognition of biochemical failure in the absence of symptoms. ADT is associated with side effects that can impact on quality of life. It is unclear whether ADT reduces prostate-specific mortality. There is currently insufficient evidence on the timing of ADT with respect to prevention of prostate cancer death and quality of life and cost particularly for men with fast and slow prostate specific antigen (PSA) doubling times.

The general objective of the ELAAT trial is to determine the optimal timing of ADT in men with recurrent prostate cancer after radical radiotherapy.

Consenting patients who have undergone prior radical radiotherapy for prostate cancer and are now experiencing a recurrence will be screened for eligibility. If they are determined to be eligible, patients will be stratified according to PSA doubling time, pre-radiation Gleason Score, previous radical prostatectomy and clinical centre. After stratification, patients will be randomized to immediate versus deferred ADT based on the 1:1 ratio between the two arms.

Patients will be followed indefinitely and assessed formally at 6 month intervals after the date or randomization. Patients will be assessed for recurrent disease (biochemical failure), new primary cancer, complications of advanced malignancy, quality of life and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Males over 18 years of age with histological confirmation of adenocarcinoma of the prostate.
2. Biochemical progression after radical radiotherapy with a total prostate dose > 52 Gy.

   * In patients without previous radical prostatectomy, biochemical progression is defined as PSA in the range of nadir + 2 ng/mL (Phoenix definition) to ≤ 6 ng/mL (this PSA must be within 30 days of randomization).
   * In patients with previous radical prostatectomy, biochemical progression is defined as a rising PSA (at least 2 values) in the range of 0.4 ng/mL to ≤ 3 ng/mL (most recent PSA must be within 30 days of randomization).

Exclusion Criteria:

1. Patients who are within 4 years of their brachytherapy implantation date.
2. Patients with medical conditions in which goserelin or bicalutamide is contraindicated in the opinion of the supervising oncologist or urologist.
3. Patients with another active malignancy or malignancy treatment within 5 years (basal or squamous cell skin cancers are not excluded from this trial).
4. Patients with geographic inaccessibility precluding them from necessary follow-up.
5. Failure to provide written informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-04; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Time to androgen independent disease (AID). AID is defined as the time from randomization to AID or last follow-up. | Every 6 months

SECONDARY OUTCOMES:
Time to complications of advanced malignancy (CAM) and number of CAMs experienced are secondary outcome measures. | Every 6 months
  The time to CAM will be defined as the interval from randomization to the first CAM.
Quality of life | Every 6 months
  Measured at each 6 - month follow-up visit using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC).
Cause Specific Survival. | Every 6 months
  The following will be considered as endpoints in assessing cause-specific survival: (1) Death adjudicated as due to prostate cancer (2) Death due to complications of ADT, irrespective of the status of malignancy.
Overall survival | Every 6 months
  Defined as the time from randomization to the time of death (from any cause) or to the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Loblaw, MD, Principal Investigator — Odette Cancer Centre - Sunnybrook Health Sciences Centre
Locations (11):
- Canada (11):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Odette Cancer Centre - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - CHUM - Hôpital Notre-Dame, Montreal, Quebec
  - McGill Clinical Research Program, Montreal, Quebec
  - CHUQ, L'Hotel-Dieu de Quebec, Québec, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan